CLINICAL TRIAL: NCT07259902
Title: Mapping the Neuroplasticity of Patients Affected by Chronic Temporomandibular Disorders on fMRI
Brief Title: FMRI Study on DC/TMD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Marco Farronato, CO-Principal Investigator, University of Milan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DC/TMD01
Record Dates: First submitted 2025-09-30; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): FMRI
  Interventions: Diagnostic Test: fMRI
- Healthy controls (Active Comparator): FMRI
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — fMRI morphological analysis

SUMMARY:
Temporomandibular disorders (TMD) are among the most common causes of chronic pain worldwide. It is estimated that about 5-12% of the global population is affected, and some conditions, such as arthritis, may be causative factors. Depending on severity, the joints involved can affect multiple functions of the masticatory system, such as the ability to speak, chew, swallow, limit facial expressions, and even breathe. Moreover, most patients with TMD may report painful conditions in other parts of the body, with comorbidities including chronic fatigue syndrome, chronic headache, endometriosis, fibromyalgia, interstitial cystitis, irritable bowel syndrome, back pain, sleep disorders, and vulvodynia. Another significant condition that frequently occurs alongside TMD is psychological distress in the form of anxiety and/or depression.

The study proposed by this research protocol aims to investigate the presence of TMD and associated psychological/psychiatric disorders such as anxiety and depression. The innovative value of the research lies in evaluating whether the association between these disorders may lead to neuroplastic changes at the brain level, which could guide targeted therapies. Only a few studies in the literature have explored this possible association, with inconclusive and conflicting results.

The study will be prospective in design, based on reference clinical/diagnostic criteria and functional neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Afflicted with temporomandibular disorder (TMD) associated with chronic pain diagnosed by an experienced specialist among the authors; the disorder, to be considered chronic, must have been present for at least six months.
* Patients with adequate sensorimotor abilities to participate in the study. This included sufficient vision to read from a computer or tablet screen at a normal distance, sufficient hearing ability to understand normal language, and sufficient motor ability to control a table mouse or computer.

Exclusion Criteria:

* Control subjects, participating voluntarily in the study, must have met the following inclusion criteria:
* Healthy subjects defined as free from temporomandibular disorders or diagnosed psychological and/or psychiatric disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
fmri Blood Oxygen Level-Dependent (BOLD) | end of the fmri
  Oxygenation concentration (referred to as BOLD). Bold is primarily used on the other hand to conduct function brain mapping. The degree of BOLD is a measure of the neuronal activity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided